CLINICAL TRIAL: NCT06873087
Title: Alterations in PACAP, CGRP, and VIP Levels in Rosacea Patients Receiving Systemic Isotretinoin Treatment: Association with Erythema Index
Brief Title: Changes in PACAP, CGRP, and VIP Levels in Rosacea Patients on Systemic Isotretinoin and Their Association with Erythema
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: SB Istanbul Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yusuf Mert Döş, Principal investigator, SB Istanbul Education and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBIstanbul_YMD
Record Dates: First submitted 2025-03-01; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Rosacea
Keywords: rosacea; isotretinoin; cgrp; vip; pacap; erythema index
MeSH Terms: conditions — Rosacea | interventions — Isotretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Rosacea patients (Other): Patients with neuropeptide values calculated before and after isotretinoin treatment
  Interventions: Drug: İsotretinoin

INTERVENTIONS:
Drug: İsotretinoin — Isotretinoin treatment at a dose of 0.3 mg/kg/day for 3 months

SUMMARY:
The goal of this clinical study is to investigate the effects of systemic isotretinoin on vasoactive neuropeptides (PACAP, VIP, CGRP) and its relationship with the erythema index in patients with rosacea. It also aims to assess the clinical efficacy of isotretinoin in reducing rosacea severity. The main questions this study seeks to answer are:

Does systemic isotretinoin treatment lead to changes in PACAP, VIP, and CGRP levels in rosacea patients? How does isotretinoin affect erythema and overall rosacea severity? Researchers will compare pre- and post-treatment neuropeptide levels and erythema index measurements to determine the effects of isotretinoin.

Participants will:

Take 0.3 mg/kg/day of isotretinoin for three months Undergo monthly clinical evaluations with RASI and erythema index measurements Have blood samples collected at baseline and after treatment to assess changes in PACAP, VIP, and CGRP levels

DETAILED DESCRIPTION:
This clinical study investigates the effects of systemic isotretinoin on vasoactive neuropeptides (PACAP, VIP, CGRP) and its relationship with erythema severity in rosacea patients. The study aims to explore the potential role of these neuropeptides in rosacea pathogenesis and assess isotretinoin's impact beyond its known effects on papulopustular lesions.

A total of 30 patients with papulopustular rosacea (PPR) and 35 healthy controls are included in the study. Participants are evaluated before treatment and at the 1st, 2nd, and 3rd months of isotretinoin therapy. Lesion severity is assessed using the Rosacea Area and Severity Index (RASI), while erythema is objectively measured with a Mexameter device. Blood samples are collected at baseline and after three months of treatment to determine PACAP, VIP, and CGRP levels.

The study is designed to provide an objective assessment of neuropeptide levels in relation to erythema severity in rosacea and to explore potential mechanisms underlying isotretinoin's effects. Findings from this research may contribute to further investigations into VIP-targeted therapeutic strategies for erythema management in rosacea.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 75 years with a diagnosis of papulopustular rosacea (PPR)
* No history of systemic or topical medication use for rosacea or other dermatological conditions in the past four weeks
* No known autoimmune or dysregulated systemic disease
* No history of migraine, inflammatory bowel disease or malignancy
* No daily sun exposure exceeding three hours
* No excessive spice consumption (more than three times per week)
* Non-smokers
* No excessive tea or coffee consumption (more than three times per week)
* Non-alcohol consumers
* No contraindications for systemic isotretinoin treatment

Exclusion Criteria:

* Patients younger than 18 or older than 75 years or without a diagnosis of papulopustular rosacea (PPR)
* History of systemic or topical medication use for rosacea or other dermatological conditions in the past four weeks
* Presence of a known autoimmune or dysregulated systemic disease
* History of migraine, inflammatory bowel disease, or malignancy
* Daily sun exposure exceeding three hours
* Frequent spice consumption (more than three times per week)
* Smokers
* Excessive tea or coffee consumption (more than three times per week)
* Alcohol consumers
* Presence of contraindications for systemic isotretinoin treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in PACAP Levels in Rosacea Patients at the End of the 3-Month Systemic Isotretinoin Treatment | Baseline and at the end of the 3-month systemic isotretinoin treatment.
  This study examines the change in PACAP levels in rosacea patients at the end of a 3-month systemic isotretinoin treatment. Blood samples are collected at baseline and after 3 months of treatment to assess the potential effects of isotretinoin on PACAP regulation. The study aims to explore the role of PACAP in the pathogenesis of rosacea and evaluate whether isotretinoin influences its expression in circulation.
Change in CGRP Levels in Rosacea Patients at the End of the 3-Month Systemic Isotretinoin Treatment | Baseline and at the end of the 3-month systemic isotretinoin treatment.
  This study examines the change in CGRP levels in rosacea patients at the end of a 3-month systemic isotretinoin treatment. Blood samples are collected at baseline and after 3 months of treatment to assess the potential effects of isotretinoin on CGRP regulation. The study aims to explore the role of CGRP in the pathogenesis of rosacea and evaluate whether isotretinoin influences its expression in circulation.
Change in VIP Levels in Rosacea Patients at the End of the 3-Month Systemic Isotretinoin Treatment | Baseline and at the end of the 3-month systemic isotretinoin treatment.
  This study examines the change in VIP levels in rosacea patients at the end of a 3-month systemic isotretinoin treatment. Blood samples are collected at baseline and after 3 months of treatment to assess the potential effects of isotretinoin on VIP regulation. The study aims to explore the role of VIP in the pathogenesis of rosacea and evaluate whether isotretinoin influences its expression in circulation.

SECONDARY OUTCOMES:
Change in Rosacea Area and Severity Index (RASI) throughout the 3-month systemic isotretinoin treatment | Baseline, 1st month, 2nd month, and 3rd month of systemic isotretinoin treatment. ( 12 weeks)
  This study evaluates the Rosacea Area and Severity Index (RASI) change throughout a 3-month systemic isotretinoin treatment in patients with papulopustular rosacea (PPR). RASI scores are assessed at baseline and at the first, second, and third months of treatment to monitor the progression of lesion severity over time. The study aims to provide objective data on isotretinoin's efficacy in reducing rosacea severity and to explore its potential effects beyond papulopustular lesions.
Change in Erythema Index throughout the 3-month systemic isotretinoin treatment | Baseline, 1st month, 2nd month, and 3rd month of systemic isotretinoin treatment. ( 12 weeks)
  This study investigates the Erythema Index (EI) change throughout a 3-month systemic isotretinoin treatment in patients with papulopustular rosacea (PPR). EI measurements are taken at baseline, 1st, 2nd, and 3rd months using a Mexameter device to assess erythema severity over time. The study aims to evaluate the impact of isotretinoin on erythema and explore its potential effects on vascular and inflammatory responses in rosacea.

CONTACTS AND LOCATIONS:
Overall Officials: yusuf m döş, MD, Principal Investigator — Istanbul Training and Research Hospital
Locations (1):
- Istanbul Training and Research Hospital, Istanbul, fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR